CLINICAL TRIAL: NCT07094399
Title: Tranexamic Acid for Postpartum Vaginal Laceration Hemorrhage
Status: Completed | Type: Observational
Sponsor: Harran University (Other)
Collaborators: Esra Söylemez, MD (Mardin Education and Research Hospital) (Unknown); Emre Uysal, MD (Yusufeli State Hospital) (Unknown)
Responsible Party: Principal Investigator, Omer Tammo, MD, Principal Investigator, Harran University
Other Study IDs: HRÜ/24.20.49
Record Dates: First submitted 2025-06-03; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Postpartum Hemorrhage; Vaginal Lacerations
Keywords: Postpartum hemorrhage; vaginal laceration; tranexamic acid; topical administration; intravenous administration.
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The necessary information was provided to the patients included in the study and their written consent was obtained.

DETAILED DESCRIPTION:
Study Design:

This study was conducted as a prospective, randomized controlled trial at the Department of Obstetrics and Gynecology of Mardin Training and Research Hospital between January 2024 and November 2024.

Participants:

A total of 161 women meeting the inclusion criteria were enrolled in the study. Inclusion criteria were:

* Vaginal delivery without episiotomy
* Presence of superficial vaginal lacerations
* Postpartum blood loss not exceeding 500 ml
* Age between 20 and 35 years
* Informed consent obtained

Exclusion criteria were:

* Cesarean delivery
* Episiotomy or vaginal lacerations requiring suturing
* Postpartum bleeding exceeding 500 ml
* Pre-existing coagulation disorders
* Tranexamic acid allergy

Randomization and Group Allocation:

Eligible participants were randomly assigned in a 1:1:1 ratio to one of three groups using a computer-generated random number sequence. The randomization sequence was generated using SPSS software version 20.0 (IBM Corp., Armonk, NY, USA). To ensure allocation concealment, the randomization sequence was kept in sequentially numbered, sealed envelopes. Envelopes were opened only after the participant had provided informed consent and was confirmed to be eligible by a researcher not involved in the treatment administration.

* Topical Tranexamic Acid Group (n=54): Received topical tranexamic acid.
* Intravenous Tranexamic Acid Group (n=54): Received intravenous tranexamic acid.
* Control Group (n=53): Received standard postpartum care without tranexamic acid.

Interventions:

* Topical Tranexamic Acid Group:

  * A sterile gauze compress (10x10 cm) was soaked with 1 gram of tranexamic acid (TXA) in 10 ml of sterile saline solution.
  * The TXA solution was prepared by diluting 10 ml of TXA (100mg/ml) in 10 ml of sterile saline.
  * The vaginal laceration(s) were assessed for length and depth using a sterile ruler prior to application.
  * The gauze was folded to ensure it covered the entire lacerated area.
  * Sterile retractors were used to gently separate the vaginal walls and ensure direct contact of the gauze with the laceration(s) while avoiding contact with the vaginal walls.
  * The retractors were held in place for 10 minutes.
  * After 10 minutes, the gauze and retractors were removed, and the area was gently washed with 20 ml of sterile physiological saline.
* Intravenous Tranexamic Acid Group:

  * 1 gram of tranexamic acid (1 gram/10 cc) was diluted in 100 ml of 0.9% NaCl isotonic solution.
  * The TXA solution was infused intravenously over 10 minutes via a peripheral venous catheter in the antecubital fossa.
  * The infusion rate was set at 100 mg/min.
  * After the infusion, the line was flushed with 5 ml of 0.9% NaCl isotonic solution.
* Control Group:

  * Participants in the control group received standard postpartum care, which included observation and monitoring of bleeding, but no tranexamic acid administration.
  * If bleeding persisted or worsened, standard institutional protocols for PPH management were followed, which may have included uterotonics, manual removal of clots, or further interventions as deemed necessary by the attending physician.

Standard Postpartum Care:

All participants received standard postpartum care according to the hospital's protocol, which included:

* Uterine massage every 15 minutes for the first hour
* Monitoring of vital signs (blood pressure, heart rate) every 15 minutes for the first hour and then hourly
* Assessment of fundal height and uterine tone every 15 minutes for the first hour and then hourly
* Perineal care with sterile pads
* Regular assessment of vaginal bleeding

Outcome Measures:

The primary outcome was the total amount of postpartum blood loss within the first 3 hours after delivery, measured using the gravimetric method.

Secondary outcomes included:

* Number of pads used in the first 3 hours postpartum
* Change in hemoglobin, hematocrit, and platelet counts from before delivery to 3 hours postpartum
* INR values before delivery and 3 hours postpartum
* Length of hospital stay (hours)
* Occurrence of complications (e.g., infection, hematoma, allergic reaction)

Blood Loss Measurement:

Postpartum blood loss was measured using the gravimetric method. All perineal pads used by the participants in the first 3 hours after delivery were collected and weighed. The dry weight of each pad was recorded before use using a calibrated digital scale with 1 gram sensitivity. After use, the wet weight of each pad was measured immediately after removal. The difference between the wet and dry weight was assumed to be the amount of blood loss, with 1 gram of weight gain considered equivalent to 1 ml of blood loss. The total blood loss was calculated by summing the blood loss from all pads used by each participant.

Laboratory Measurements:

Hemoglobin (Hb), hematocrit (Hct), platelet counts, and INR values were measured from venous blood samples taken before delivery (within 1 hour before delivery) and at the 3rd hour postpartum. Blood samples were collected in standard EDTA and citrate tubes and analyzed at the hospital's central laboratory using standard laboratory procedures.

Sample Size Calculation:

The sample size was calculated using G*Power software (version 3.1.9.2, Universität Kiel, Germany). Based on a previous study [cite a similar study if possible, provide details], with an estimated effect size of 0.6 for the primary outcome (blood loss), an alpha level of 0.05, and a desired power of 80%, the calculated minimum sample size required was 50 patients per group. To account for potential dropouts and ensure adequate power, we aimed to recruit 54 patients per group.

ELIGIBILITY:
Study Population: 161 women aged 20-35 years who had spontaneous vaginal deliveries.

Sampling Method: Non-Probability Sample

Minimum Age: 20 Years

Maximum Age: 35 Years

Sex: Female

Gender Based: Yes

Accepts Healthy Volunteers: Yes

Criteria:

Inclusion Criteria:

Vaginal delivery without episiotomy

Presence of superficial vaginal lacerations

Postpartum blood loss not exceeding 500 ml

Age between 20 and 35 years

Informed consent obtained

Exclusion Criteria:

Cesarean delivery

Episiotomy or vaginal lacerations requiring suturing

Postpartum bleeding exceeding 500 ml

Pre-existing coagulation disorders

Tranexamic acid allergy

-

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — MALE
Study Population: 161 women aged 20-35 years who had spontaneous vaginal deliveries.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Total Postpartum Blood Loss | Within the first 3 hours after delivery
  The total amount of postpartum blood loss within the first 3 hours after delivery, measured using the gravimetric method by weighing blood-soaked pads. The difference between the wet and dry weight of the pads was assumed to be the amount of blood loss, with 1 gram of weight gain considered equivalent to 1 ml of blood loss.

SECONDARY OUTCOMES:
Number of Pads Used | First 3 hours postpartum
  The count of perineal pads used by participants within the first 3 hours postpartum to assess blood loss.

OTHER OUTCOMES:
Change in Hemoglobin (Hb) Levels | Before delivery (within 1 hour before delivery) and at 3 hours postpartum.
  Change in hemoglobin levels, measured from venous blood samples. Unit of Measure: g/dL (grams per deciliter).
INR Values | Before delivery and at 3 hours postpartum
  International Normalized Ratio (INR) values were measured from venous blood samples.
Change in Hematocrit (Hct) Levels | Time Frame: Before delivery (within 1 hour before delivery) and at 3 hours postpartum. Unit of Measure: % (percentage).
  Change in hematocrit levels, measured from venous blood samples.
Length of Hospital Stay | From birth until discharge, typically 1 to 4 days postpartum, as measured in this study.
  The total duration of hospital stay for participants following vaginal delivery.
Incidence of Complications | From birth until hospital discharge, within an average of 1 to 4 days postpartum
  The occurrence of complications, including infection, hematoma, or allergic reaction, observed in participants.
Change in Platelet (PLT) Counts | Before delivery (within 1 hour before delivery) and at 3 hours postpartum.
  Change in platelet counts, measured from venous blood samples.Unit of Measure:Unit of Measure: ×10 3 /μL (cells per microliter)

CONTACTS AND LOCATIONS:
Overall Officials: ömer tammo, Study Director — omertammo@harran.edu.tr
Locations (1):
- Harran University, Sanliurfa, Şanliurfa, Turkey (Türkiye)

REFERENCES:
- [Derived] Tammo O, Uysal E. Effectiveness of tranexamic acid in intervening postpartum vaginal lacerations. BMC Pregnancy Childbirth. 2025 Dec 16. doi: 10.1186/s12884-025-08584-y. Online ahead of print. PMID 41398944